CLINICAL TRIAL: NCT01845467
Title: Efficacy of Secretin Assisted Dynamic MRCP in the Diagnosis and Follow up of Auto Immune Pancreatitis(AIP)
Brief Title: Efficacy of Secretin MRCP in the Diagnosis and Follow up of Auto Immune Pancreatitis
Acronym: S-MRCP
Status: Withdrawn | Type: Observational
Why Stopped: Unable to enroll participants
Sponsor: Johns Hopkins University (Other)
Collaborators: ChiRhoClin, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NA_00068830
Record Dates: First submitted 2013-04-15; First posted 2013-05-03 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Cellular Diagnosis, Pancreatic Cancer; Autoimmune Pancreatitis
Keywords: Secretin MRCP, diagnosis, Autoimmune pancreatitis
MeSH Terms: conditions — Pancreatic Neoplasms; Autoimmune Pancreatitis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Auto-immune pancreatitis, suspected: Patients suspected with auto-immune pancreatitis (AIP) and undergoing secretin assisted MRCP as per the standard of care at our institute.

SUMMARY:
BACKGROUND:

Auto immune pancreatitis (AIP), a benign pancreatic disease has certain morphological forms which mimics pancreatic malignancy in radiological appearance. There is no singe diagnostic test which can accurately differentiate these two conditions. In the past, AIP accounted for up to 27% of Whipple resections performed for suspected adenocarcinoma.

AIMS:

To evaluate the efficacy of Secretin assisted Magnetic resonance cholangio pancreatography (MRCP) in differentiating AIP and pancreatic malignancy.

METHODS:

100 patients suspected with AIP will be consented to participate in the study to undergo secretin MRCP in addition to their other standard investigations. Patients will be categorized as those with AIP and with pancreatic malignancy based on these results and will be followed. Follow up will eventually give the true diagnosis when patients with pancreatic malignancy undergo pancreatic surgery and their pancreatic tissue is examined by histopathologist. AIP patients will undergo steroid trial which will give the true diagnosis. The preliminary diagnosis results based on standard investigations with and without inclusion of secretin MRCP will be compared to the true diagnosis.

DETAILED DESCRIPTION:
A total of 100 patients with suspicion of Auto Immune Pancreatitis will be identified from the multidisciplinary pancreatic cancer clinic at Johns Hopkins and from the Pancreatitis clinic of the Division of Gastroenterology, Johns Hopkins Hospital.

After written, informed consent is obtained; preliminary screening will be done which includes medical history and physical examination including weight and vital signs. Serum immunoglobulin G4 (IgG4) levels will also be evaluated. If the patient meets exclusion/inclusion criteria, screening eligibility and signs informed consent, they will be included in the study.

Study investigators and/or their delegate will complete the patient demographic form, medical history form, baseline physical examination, baseline laboratory evaluation and concomitant medication evaluation as per the protocol. Any other investigational procedure such as endoscopic ultrasonography - fine-needle aspiration (EUS - FNA) or esophagogastroduodenoscopy (EGD) with papillary biopsy for IgG4 which assists in the differentiation between AIP and Pancreatic malignancy may be performed based on the treating physician's discretion.

Involvement of other organs by AIP and Pancreatic malignancy will be obtained based on the medical history, examination and imaging findings. The patients will be subjected to MRI and MRCP with the MRCP performed in two stages namely before injection of secretin and after intravenous injection of 0.4mcg/Kg of synthetic human secretin (CHIROSTIM, Human Secretin, CHIRHOCLIN Inc., Burtonsville, MD). All the subjects will be given 3 cups (approximately 500-600cc) of pineapple juice 5-10 minutes before the imaging procedure. Pineapple juice will act as a negative oral contrast which nulls the signal in stomach and duodenum, thereby suppressing gastrointestinal overlap over pancreas. MR Examination will be performed using 3.0 T magnet and it will include non contrast enhanced scanning followed by gadolinium enhanced scanning, performed during the arterial dominant, venous dominant and late phases. The secretin MRCP is performed through serial breath-hold T2-weighted sequences run during the first 8-12 min after the intravenous administration of secretin.

Based on the result from the above investigations, the patients will be categorized as those suspected with AIP and those suspected with Pancreatic malignancy. Patients with suspected malignancy will eventually undergo surgical resection of pancreas under their treating physician and the pancreatic tissue examination will provide the true diagnosis. Patients with suspected AIP will undergo a steroid trial for at least 3 months, at the end of which a repeat MRI, secretin MRCP will be performed and the diagnosis will be confirmed based on the response to steroid therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >18 years of age.
2. Patients suspected of having AIP based on prior clinical work up

Exclusion Criteria:

1. Unwilling or unable to give written, informed consent.
2. Presence of pace makers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body.
3. Patients with acute pancreatitis

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 100 patients with suspicion of Auto Immune Pancreatitis will be identified from the multidisciplinary pancreatic cancer clinic at Johns Hopkins and from the Pancreatitis clinic of the Division of Gastroenterology, Johns Hopkins Hospital. The patients will be managed as part of standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Evaluating the additive benefit of Secretin MRCP in differentiating focal AIP and Pancreatic malignancy | Participants will be followed during the interval between initial S MRCP and a repeat S MRCP after steroid treatment or a pancreatic surgery; an expected 4 weeks
  Patients with suspected auto-immune pancreatitis (AIP)will undergo secretin assisted MRCP. The MRCP will be evaluated for post secretin changes in pancreatic dimensions, duodenal filling, pre and post contrast parenchymal signal intensities, ADC values, changes in pancreatic duct strictures due to secretin, extra pancreatic lesions.

SECONDARY OUTCOMES:
Efficacy of Secretin MRCP in monitoring therapeutic improvement in AIP patients on steroid trial | Participants will be followed up from initial S MRCP till resolution of pathology or till end of S MRCP follow-up studies; an expected 8 weeks
  The patients with suspected AIP based on secretin MRCP will undergo a steroid trial. The initial and follow up MRCP findings will be compared for changes in pancreatic parenchyma after injecting secretin, T1 signal intensities, ADC values, changes in pancreatic duct strictures,extra pancreatic lesions and duodenal filling.

CONTACTS AND LOCATIONS:
Overall Officials: Atif Zaheer, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kamisawa T, Egawa N, Nakajima H, Tsuruta K, Okamoto A, Kamata N. Clinical difficulties in the differentiation of autoimmune pancreatitis and pancreatic carcinoma. Am J Gastroenterol. 2003 Dec;98(12):2694-9. doi: 10.1111/j.1572-0241.2003.08775.x. PMID 14687819
- [Background] Carbognin G, Girardi V, Biasiutti C, Camera L, Manfredi R, Frulloni L, Hermans JJ, Mucelli RP. Autoimmune pancreatitis: imaging findings on contrast-enhanced MR, MRCP and dynamic secretin-enhanced MRCP. Radiol Med. 2009 Dec;114(8):1214-31. doi: 10.1007/s11547-009-0452-0. Epub 2009 Sep 30. PMID 19789959
- [Background] Chari ST, Takahashi N, Levy MJ, Smyrk TC, Clain JE, Pearson RK, Petersen BT, Topazian MA, Vege SS. A diagnostic strategy to distinguish autoimmune pancreatitis from pancreatic cancer. Clin Gastroenterol Hepatol. 2009 Oct;7(10):1097-103. doi: 10.1016/j.cgh.2009.04.020. Epub 2009 May 4. PMID 19410017